CLINICAL TRIAL: NCT01818271
Title: Phase 1 Study of the Effects of a Community-based Group Rehabilitation Program for Dynamic Balance and Mobility; as an Alternate to Out-patient Rehabilitation Post Stroke;
Brief Title: Effects of a Community-based Group Rehabilitation Program for Dynamic Balance and Mobility Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hr2013:086
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2013-03

CONDITIONS: Sequelae of Stroke
Keywords: community-stroke-rehabilitation,; group-exercise,; balance-mobility-exercise,; instrumented treadmill

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional physical Therapy (Active Comparator): will receive a conventional out-patient program which will include: lower extremity stretching and strengthening exercise; fitness using cycle ergometer; balance exercises in standing; over ground walking and stair exercises
  Interventions: Behavioral: conventional physical therapy
- community-based group rehabilitation (Experimental): Group training will include different workstations to target dynamic standing balance and walking. The key features includes facilitate repetition of task-related movements, tailored to the patient and patient's goals, in a meaningful context. Specifically:
  * Advanced dynamic tasks, including stepping and other transitional tasks to treadmill & over ground walking) with use of various inexpensive exercise "assistive" equipment such as mini-exercise stepper or elliptical machines.
  * Treadmill walking exercise program.
  Interventions: Behavioral: community-based group rehabilitation

INTERVENTIONS:
Behavioral: conventional physical therapy — will receive a conventional out-patient program which will include: lower extremity stretching and strengthening exercise; fitness using cycle ergometer; balance exercises in standing; over ground walking and stair exercises
  Arms: conventional physical Therapy
Behavioral: community-based group rehabilitation — Group training will include different workstations to target dynamic standing balance and walking. The key features includes facilitate repetition of task-related movements, tailored to the patient and patient's goals, in a meaningful context. Specifically:
  * Advanced dynamic tasks, including stepping and other transitional tasks to treadmill & over ground walking) with use of various inexpensive exercise "assistive" equipment such as mini-exercise stepper or elliptical machines.
  * Treadmill walking exercise program.
  Arms: community-based group rehabilitation

SUMMARY:
Stroke patients clearly benefit from intensive and coordinated inpatient care. While inpatient rehabilitation care is the preferred form for many patients post-stroke, due to access and financial barriers, many patients do not have this option. Community, outpatient rehabilitation programs will allow the patients with moderately disabling strokes the opportunity to maintain or augment gains achieved during inpatient stroke rehabilitation , while allowing some patients with mild disability to avoid inpatient rehabilitation completely.

Objective: Phase 1 randomized control trial to test the efficiency and effectiveness of treating adults who have suffered a single stroke using the following essential treatment components; a) community setting, b) group activity program, c) flexible, task-specific, computer-based exercise regime This program is designed to allow an extension of the in-patient rehabilitation experience to a community-based setting, in a cost-effective manner using paraprofessional staff and rehabilitation specialists, to provide a challenging, functional program to promote recovery and independence from physical impairments affecting balance and walking.

The specific objectives are to:

1. assess the benefits and feasibility of the multi-functional group exercise intervention for balance and mobility in a community setting. Secondary objectives
2. identify effective combinations of exercises & activities that translate to increased abilities and participation levels.

Hypothesis: Intense training targeting standing balance, and walking will significantly improve stroke clients' functional mobility. Training in a group setting and incorporating interactive and engaging computer gaming further provides the benefits of motivation and peer support while providing treatment in a cost effective manner.

ELIGIBILITY:
Inclusion Criteria:

1. community dwelling individuals, who have suffered a single stroke of thrombic -embolic or hemorrhagic origin in the last 3-12 months and are waiting for outpatient rehabilitation ,
2. Aged 50-70 years,
3. Montreal Cognitive Assessment score greater than 26,
4. English-speaking and possess the ability to understand the nature of the study and provide informed consent,
5. Independent in sit to stand transfer and ambulatory functions, with or without an assistive device (cane or walker), f ) Gait speed (average over 25 meters) between 0.3 and 0.8 m/s and Berg Balance Scale score of less than 45.

Exclusion Criteria:

Any medical condition or disability that prevents participation in an exercise program. For example, a reported medical history of current treatment for cancer, kidney disease, recent fracture, uncontrolled diabetes or seizure disorder, uncontrolled cardiovascular-related problems .

-

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Gait speed | pre and post intervention of 8 weeks
  Proportion of participants with an improved functional level of walking As per LEAPS multi-centre RCT.47 Improved functional level was defined as; (a) the ability to walk independently at a speed of 0.8 m per second or faster for persons with initially moderate gait impairment , or (b) ability to walk independently at a speed of 0.4 m per second or faster for persons with initially severe gait impairment. These transitions are associated with improvements in home or community ambulation, functional status, and quality of life.50
Stroke Impact Scale | Pre and post intervention of 8 weeks
  This scale is a self reported, stroke specific, valid, reliable, and responsive measure that includes 59 items and assesses eight domains related to activities and participation.

SECONDARY OUTCOMES:
Berg Balance Scale | pre and post intervention of 8 weeks
Timed Up and Go Test | Pre and Post intervention of 8 weeks

OTHER OUTCOMES:
6-minute wlak test | Pre and Post intervention of 8 weeks
Spatial-Temporal gait variables | pre and post intervention of 8 weeks
  . Spatial-Temporal gait parameters using instrumented walkway.56 Average walking speed (in 4 meters) mean and variance measurement (over 20 steps) will be obtained for the following parameters: swing and stance duration, single support

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm Szturm, PT, PhD, Principal Investigator — Faculty of Medicine University of Manitoba; Sepideh Pooyania, MD, Principal Investigator — Faculty of Medicine University of Manitoba
Locations (2):
- Canada (2):
  - School of Medical Rehabilitation , University of Mantioba, Winnipeg, Manitoba
  - Riverview Health Centre, Winnipeg, Manitoba